CLINICAL TRIAL: NCT04808570
Title: A Single-arm, Open-label, Multi-center Phase Ib/II Study of TQ-B3525 in Subjects With Relapsed/Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma(CLL/SLL)
Brief Title: A Study of TQ-B3525 in Subjects With Relapsed/Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The sponsor terminated the study due to the R&D strategy change.
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQ-B3525-Ib/II-06
Record Dates: First submitted 2021-03-11; First posted 2021-03-22 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-10

CONDITIONS: Relapsed/Refractory Chronic Lymphocytic Leukemia/Small Lymphocytic Lymphoma
MeSH Terms: conditions — Recurrence | interventions — TQ-B3525

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQ-B3525 tablets (Experimental): TQ-B3525 tablet administered orally.
  Interventions: Drug: TQ-B3525 tablets

INTERVENTIONS:
Drug: TQ-B3525 tablets — TQ-B3525 tablet administered 20mg orally, once daily in 28-day cycle.

SUMMARY:
This is a study to evaluate the efficacy and safety of TQ-B3525 in subjects with relapsed/refractory chronic lymphocytic leukemia/small lymphocytic lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* 1.Understood and signed an informed consent form; 2. 18 years and older, Eastern Cooperative Oncology Group(ECOG) performance status score of 0 to 2, Life expectancy ≥ 3 months; 3.Chronic lymphocytic leukemia/small lymphocytic lymphoma diagnosed by flow cytometry or pathology, and meets at least one of the criteria for active diseases requiring treatment in IWCLL2008; 4.Has received at least one line of previous treatment, the latest treatment confirmed no objective response, or disease progress after treatment; 5.Has at least one measurable lesion; 6. Adequate organ system function; 7. Male or female subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study (such as intrauterine devices , contraceptives or condoms) ；No pregnant or breastfeeding women, and a negative pregnancy test are received within 7 days before the first administration.

Exclusion Criteria:

-1. Has Richter's transformation or prolymphocytic leukemia (PLL)； 2. Has central nervous system violation; 3. Has uncontrolled primary autoimmune cytopenias, including autoimmune hemolytic anemia (AIHA), idiopathic thrombocytopenic purpura (ITP), etc； 4. Has received other PI3K inhibitors or CAR-T treatments; 5. Has diagnosed and/or treated additional malignancy within 3 years prior to the first administration; 6.Diagnosed as type I diabetes or uncontrollable type II diabetes, or fasting blood glucose> 8.9 mmol/L or glycosylated hemoglobin (HbA1c)> 8.5% during the screening period; 7. Has interstitial lung disease or drug-induced interstitial lung disease history; 8. Has a history of immunodeficiency diseases; 9. Has multiple factors affecting oral medication; 10. Has adverse events caused by previous therapy except alopecia that did not recover to ≤grade 1; 11. Has received systemic steroid treatment within 7 days before the first administration; 12. Has received other systemic anti-tumor medications within 4 weeks before the first administration, or still within the 5 half-life of the medication, which occurs first; 13.Has active infections within 4 weeks before the first administration; 14.Has received surgery, or unhealed wounds within 4 weeks before the first administration; 15. Has a history of autologous hematopoietic stem cell transplant within 3 months; 16. Has a history of allogeneic hematopoietic stem cell transplant; 17. Grade II or higher cardiovascular disease within 6 months before the first administration; 18.QTCF > 480ms, LVEF < 50%; 19.Urinary protein ≥ 2 +, and 24-hour urinary protein quantity>1g within 7 days; 20. Has active hepatitis B or C; 21. Has psychotropic substances abuse or a mental disorder; 22. Has other conditions that make it inappropriate for the patient to be enrolled based on investigator's opinion.

21. Has psychotropic substances abuse or a mental disorder;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2021-06-05 (Actual); Primary Completion 2023-11-22 (Actual); Study Completion 2023-11-22 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) assessed by Independent Review Committee | Baseline up to 18 months
  Percentage of participants achieving complete response (CR) and partial response (PR) based on IRC

SECONDARY OUTCOMES:
Overall response rate (ORR) assessed by Investigator | Baseline up to 18 months
  Percentage of participants achieving complete response (CR) and partial response (PR) assessed by investigator.
Duration of disease remission (DOR) | Baseline up to 18 months
  The time from the first evaluation of the subject as CR or PR to the first evaluation of the subject as PD or death (whichever occurs first).
Progression-free survival (PFS) | Baseline up to 18 months
  PFS was defined as the time from the date of study enrollment to the date of the first of the following events, objective disease progression or death due to any cause
Disease control rate（DCR） | Baseline up to 18 months
  Percentage of subjects achieving complete response (CR) and partial response (PR) and stable disease (SD).
Overall Survival (OS) | Baseline up to 24 months
  OS defined as the time from the first dose to death from any cause. Survival time was censored at the date of last contact for patients who were still alive or lost to follow-up.
Incidence of Adverse Events, Serious Adverse Events | Baseline up to 18 months
  AE, SAE, and withdrawal from the trial for reasons such as safety or tolerability.

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - The First Affiliate Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Hematology Hospital of Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality